CLINICAL TRIAL: NCT05759338
Title: A Study of Revian Red All LED Cap as a Novel Treatment for Central Centrifugal Cicatricial Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00094234
Record Dates: First submitted 2023-02-24; First posted 2023-03-08 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-12

CONDITIONS: Central Centrifugal Cicatricial Alopecia
Keywords: hair loss; scalp symptoms
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Using the Revian Red All LED cap 10 minutes each day for 6 months
  Interventions: Device: Revian Red All LED cap

INTERVENTIONS:
Device: Revian Red All LED cap — The cap is a dual-band LED light therapy wireless "smart" cap. It has been shown to be effective in androgenetic alopecia (used once daily, 10-minute treatment regimen) for both men and women.

SUMMARY:
The purpose of this study is to determine if the Revian Red All LED cap shows potential to be an effective treatment for Central centrifugal cicatricial alopecia (CCCA) by recruiting hair follicles back to anagen growth or by improving inflammation. The primary outcome is to determine if hair loss regression is halted. Secondary outcomes include hair regrowth and alleviation of signs and symptoms of the disease.

Participants will be asked to use the Revian Red All LED cap once daily for a 10-minute treatment regimen which is the current androgenetic alopecia recommendation.

DETAILED DESCRIPTION:
Subjects who are willing to participate in a novel treatment for Revian Red All LED cap will be enrolled in this study. The cap uses two wavelengths of light, 620 nm and 660 nm. A study cap will be provided for each subject. Subjects will use the cap once daily, 10-minute treatment regimen which is the current androgenetic alopecia recommendation. The subjects will use the cap for a total of 6 months. To use the cap, subjects will connect the Revian Red All LED cap to a Smart App on a mobile phone device using Bluetooth. Subjects can use the Smart App to set daily reminders to use the cap, track and log usage, and use the 10 minute timer. No additional information will be stored on the Smart App. Only subjects will have access to the Smart App located on their personal mobile phone device.

Standardized photos and trichoscopic photos before starting treatment and every 2 months for x 6 total months will be taken to assess hairline stabilization and potential for regrowth. A baseline photo and completion photo will also be taken with a visio device. This will help determine pigmentation of the present hairs throughout the study.

Prior to study enrollment, all participants will receive a detailed explanation of the purpose of the study and will undergo written informed consent. Clinical history of hair loss and history of prior treatment will be obtained by administering a standardized questionnaire to all subjects. Subjects will also fill out a questionnaire regarding symptoms of their hair loss at each visit. There will be 4 visits total (1 Pre-treatment visit and 3 Follow up visits).

ELIGIBILITY:
Inclusion Criteria:

* Women who are between the age of eighteen years and sixty-five years
* Biopsy-proven diagnosis of CCCA Stage II-IV.
* Must be on stable treatment without changes (on doxycycline, topical steroids, minoxidil and/or post 8 rounds of intralesional steroids) for at least 3 months

Exclusion Criteria:

* Subjects with other forms of hair loss that is not CCCA
* Prior treatment with light source for alopecia
* Males are excluded from this study since the prevalence of CCCA in males is so significantly low that it is difficult to find cases in a clinical setting

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self identified
Enrollment: 24 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy McMichael, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 24
Completed | 21
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.79 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24
Disease Duration [Mean (Standard Deviation); unit: years] | 11.75 (8.27)

OUTCOME MEASURES:

1. Primary Outcome: Shape of the Hairline Documented With Photographs
Description: Photographs of the stabilization and regrowth of the hairline documented by standardized camera and dermatoscopic photographs of the scalp
Time Frame: Baseline to month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 21
Participants
  stabilization of hair loss | 8
  improvement in hair growth | 12
  worsened hair loss | 2

2. Secondary Outcome: Change in Hairline Assessment Scores by Participant
Description: Subjects will complete the standardized questionnaire regarding symptoms of their hair loss: Perception Dermatology Life Quality Index (DLQI) survey - The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Time Frame: Baseline to month 6
Population: Secondary outcome (Alleviation of signs and symptoms of disease):
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 21
Participants
  Improvement in symptoms: | 11
  Worsened symptoms | 6
  • Stable symptoms | 4

3. Secondary Outcome: Change in Perifollicular Scale Assessments of Hairline Change by Study Physician
Description: Scalp and hair exam and assessment with completion of grader survey to measure: Perifollicular scale
  Mild - affecting <10% of scalp. Moderate - affecting 10-30% of scalp. Severe - affecting >30% of scalp. For all signs other than Vellus/Intermediate/Terminal hair shafts: Percentage of types of hair shafts
Time Frame: Baseline to month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 21
Participants
  Improvement on trichoscopy: had a decrease in inflammatory signs | 13
  Combination of findings: Decrease in perifollicular scale | 6
  Combination of findings: Decrease in perifollicular hyperpigmentation and erythema | 13
  Combination of findings: Increased vellus hairs | 8
  Combination of findings: Decrease in disrupted honeycomb pigment network | 1
  Worsened disease on trichoscopy: Worsening perifollicular scale | 1
  Worsened disease on trichoscopy: Worsened erythema | 2
  Stable disease on trichoscopy: | 6

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT05759338/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT05759338/ICF_000.pdf